CLINICAL TRIAL: NCT03174769
Title: Effects of Higher Consumption of Protein-rich Animal Foods With the USDA Healthy U.S.-Style Eating Pattern on Sleep Quality and Cardio-metabolic Health in Overweight/Obese Adults During Diet-induced Weight Loss
Brief Title: Impact of Protein Quantity Within the USDA Healthy Style Eating Pattern on Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Principal Investigator, Purdue University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1701018623
Record Dates: First submitted 2017-05-31; First posted 2017-06-02 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Sleep; Body Composition

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Protein with weight loss (Active Comparator): weight loss subjects will consume a 750 reduced calorie daily diet based on current ht. wt and age
  Meal Pattern USDA Healthy U.S.-Style Eating Pattern with ~5 oz eq of protein foods for 12 wk
  Interventions: Other: Normal protein
- High protein and weight loss (Experimental): weight loss subjects will consume a 750 reduced calorie daily diet based on current ht. wt and age
  Meal Pattern USDA Healthy U.S.-Style Eating Pattern with ~12.5 oz eq of protein foods for 12 wk
  Interventions: Other: High protien

INTERVENTIONS:
Other: Normal protein — Following a two week baseline assessment period, subjects will consume a diet with normal protein diet while undergoing weight loss for 12 wk.
  Arms: Normal Protein with weight loss
Other: High protien — Following a two week baseline assessment period, subjects will consume a diet with high protein diet while undergoing weight loss for 12 wk.
  Arms: High protein and weight loss

SUMMARY:
This evaluates the affect of protein quantity on indices of sleep. Half the participants will be prescribed protein in the amount consistent with the USDA healthy style eating pattern, while the other half will be prescribed a diet containing 12.5 oz eq of protein.

DETAILED DESCRIPTION:
According to the National Sleep Foundation, 13% of U.S. adults were reported to sleep 6 hours or less per weeknight in 2001. Eight years later, the number increased to 20%. Also, the proportion of people experiencing a sleep problem (e.g. difficulties in initiating or maintaining sleep) several nights per week has increased dramatically (from 51% to 64% in 2001 to 2009). Getting enough and good quality sleep is essential to health. Indices of sleep, including duration, quality, and patterning are related to obesity, type 2 diabetes, cardiovascular disease, hypertension, worsen lipid-lipoprotein status, and premature death. All of these morbidities and mortality are also impacted by diet .

The 2015 Dietary Guidelines Advisory Committee recognized "an insufficient body of evidence" in the "emerging area" of "associations between sleep patterns, dietary intakes, and obesity risk" and that "a paucity of research exists on the potential impact of diet on sleep-related outcomes". Currently the majority of research has assessed the influence of sleep on energy balance or dietary choices. The reversed relation, how diet influence sleep, received much less attention. In general, diet-induced weight loss is considered to improve sleep quality and increase sleep duration. However, emerging research brings into question the impact of the macronutrient distribution during dietary energy restriction (ER) on indices of sleep. Dietary protein, due to its ability to provide tryptophan and tyrosine (precursors of neurotransmitters melatonin and dopamine), may influence sleep. Despite the fact that both diet and sleep predict obesity and chronic diseases, limited research exists on the effects of dietary energy and macronutrients, especially high-quality protein intake, on indices of sleep.

The primary aim is to assess the effects of the USDA Healthy U.S.-Style Eating Pattern with higher amounts of animal-based protein-rich foods (lean meats and eggs) on health outcomes including sleep and blood pressure.

This is a 16-week randomized, parallel, placebo-controlled, single-blind study. During baseline, participant's diet, general health, and sleep quality will be assessed. Participants will then be randomized and assigned to either the normal protein or high protein (5 vs. 12.5 oz-eq of protein foods daily) for the 12-week weight loss intervention with the energy-restriction (750 kcal/day dietary energy deficits).

ELIGIBILITY:
Inclusion Criteria:

* Male or female; age 35-65 y; BMI 25-39 kg∙m-2; weight stable (± 3 kg) 3 months pre-study; no acute illness; not diabetic; not pregnant or lactating; not currently (or within 3 months pre-study) following an exercise or weight loss program; non-smoking; not lactose intolerant; natural waist circumference ≥ 102 cm for men and ≥ 88 cm for women; fasting glucose < 110 mg/dL, systolic and diastolic blood pressures < 140/90 mmHg; serum total cholesterol < 260 mg/dL; LDL-cholesterol < 160 mg/dL; triacylglycerol < 400 mg/dL; PSQI score ≥ 5; and clinically normal serum albumin and pre-albumin concentrations. In addition, subjects who have been diagnosed by their doctor with moderate to severe sleep apnea or insomnia will be excluded during screening.

Exclusion Criteria:

* Diabetic, smoker

Ages: 35 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Disordered sleep | 12 weeks
  Will be assessed using the Actiwatch. Each participant will wear the Actiwatch on their wrist for 7 days as directed by the study coordinator. Outcome measurements include: real sleep time, latency, efficiency, wake time, and wake bouts.
Physiologic sleep onset | 12 weeks
  All participants will be given saliva collection tubes and instruction on how to collect will be in the kit given. This for our lab to measure saliva melatonin concentrations during the 7 days they are wearing the Actiwatch. Subjects will collect saliva hourly from 5 hours before to 2 hours before usual sleep time, then every 30 minutes until 1 hour before usual sleep time. Subjects will be given collections tubes and detailed collection instructions prior to the testing period. After sample collection, you will place the saliva filled tubes in there protective container and place the container in your refrigerator. You will keep collected samples until testing for that period is complete and you return them to the study coordinator (≤ 7 days).
Subjective sleep quality | 12 weeks
  Will be assessed using the Pittsburgh Sleep Quality Index questionnaire on a single testing day. The PSQI questionnaire is a clinical sleep behavior questionnaire validated for use in patients with insomnia, cancer, Parkinson's disease, and the general population. It is designed to assess indices of sleep during the preceding one-month interval and contains 19 questions using Likert scales from 0-3. All questions are categorized into seven sub-parameters (duration of sleep, sleep disturbance, sleep latency, day dysfunction due to sleepiness, sleep efficiency, subjective sleep quality, and use of sleeping medication). Each of these seven parameters is scored between 0 and 3 arbitrary units (au), which generates a summed total score of 0 to 21 au. This total score (GSS) of >5 au indicates poor sleep condition. Thus, a lower GSS score indicates better sleep condition. The PSQI also has questions that generate routine sleep duration in hours.

SECONDARY OUTCOMES:
Fasting state blood analyses | 12 weeks
  clinical blood chemistries
Blood pressure | 12 weeks
  24 h and clinical blood pressures
Body composition | 12 weeks
  BodPod

CONTACTS AND LOCATIONS:
Overall Officials: Wayne W Campbell, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hudson JL, Zhou J, Campbell WW. Adults Who Are Overweight or Obese and Consuming an Energy-Restricted Healthy US-Style Eating Pattern at Either the Recommended or a Higher Protein Quantity Perceive a Shift from "Poor" to "Good" Sleep: A Randomized Controlled Trial. J Nutr. 2020 Dec 10;150(12):3216-3223. doi: 10.1093/jn/nxaa302. PMID 33096550